CLINICAL TRIAL: NCT00242918
Title: Phase II Trial of Neoadjuvant Docetaxel and ZD 1839 (Iressa) Followed by Radical Prostatectomy in Patients With High Risk, Locally Advanced Prostate Cancer
Brief Title: Safety and Effectiveness Study of Docetaxel and ZD1839 Followed by Removal of the Prostate to Treat Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Collaborators: AstraZeneca (Industry); Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRI 8847; GIA #16134; 1839US/290; IIT# 16134
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2006-06

CONDITIONS: Prostate Cancer
Keywords: High risk; adenocarcinoma; prostate cancer; neoadjuvant
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Docetaxel; Gefitinib

INTERVENTIONS:
Drug: docetaxel
Drug: ZD1839

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the combination of docetaxel and ZD1839 on destroying prostate cancer before removal of the prostate.

DETAILED DESCRIPTION:
It is recognized that there is a subset of patients who are at high risk for progression despite aggressive treatment of localized disease at the time of detection. The critical issue is in addressing micrometastatic disease that has already developed prior to diagnosis. This study utilizes daily doses of ZD1839 and weekly docetaxel for two cycles prior to radical prostatectomy.

ZD1839 has demonstrated antiproliferative activity against human tumor xenografts and in coadministration with cytotoxic agents against prostate cell lines (PC-3 and TSU-PRI). The combination of ZD1839 and docetaxel has been reported to be feasible with an acceptable toxicity profile.

This phase II, single center trial is specifically targeting those patients with high-risk adenosarcoma of the prostate.

ELIGIBILITY:
Inclusion Criteria:

* prostate carcinoma: clinical stage T2b-3 or serum PSA>20 ng/ml or Gleason sum score 8-10.
* clinical T2 patients are eligible if endorectal coil MRI shows T3 disease, or Gleason 4+3 cancer in 5 or more biopsies (minimum of 10 biopsies total required)
* ECOG performance status of 0, 1 or 2
* adequate hematological, liver and renal function
* existing peripheral neuropathy < grade 1
* ability to tolerate oral medications.

Exclusion Criteria:

* Concurrent or prior treatment with radiation, cytotoxic, biologic therapy for prostate cancer
* any major surgery within four weeks
* prior hormonal therapy (except finasteride for obstructive voiding symptoms- -evidence of metastatic disease, confirmed by physical examination, computed tomography of the abdomen and pelvis within 45 days and by bone scan within 60 days of signing informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29
Dates: Start 2003-05; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the combination of docetaxel and ZD1839 on pathologic complete response (pCR) in radical prostatectomy specimens. Pathological complete response is defined as no microscopic evidence of neoplastic cells in the resected specimen.

SECONDARY OUTCOMES:
Evaluate the toxicity of docetaxel and ZD1839 in patients with high risk, locally advanced prostate carcinoma prior to surgical resection
Clinical Response
Assessment of margin of positivity at surgical resection
Evaluate PSA response from baseline and post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Vuky, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Greenlee RT, Hill-Harmon MB, Murray T, Thun M. Cancer statistics, 2001. CA Cancer J Clin. 2001 Jan-Feb;51(1):15-36. doi: 10.3322/canjclin.51.1.15. PMID 11577478
- [Background] Oh WK, George DJ, Kaufman DS, Moss K, Smith MR, Richie JP, Kantoff PW. Neoadjuvant docetaxel followed by radical prostatectomy in patients with high-risk localized prostate cancer: a preliminary report. Semin Oncol. 2001 Aug;28(4 Suppl 15):40-4. doi: 10.1016/s0093-7754(01)90153-8. PMID 11685727
- [Background] Dreicer R, Klein EA. Preliminary observations of single-agent docetaxel as neoadjuvant therapy for locally advanced prostate cancer. Semin Oncol. 2001 Aug;28(4 Suppl 15):45-8. doi: 10.1016/s0093-7754(01)90154-x. PMID 11685728
- [Background] Pienta KJ. Preclinical mechanisms of action of docetaxel and docetaxel combinations in prostate cancer. Semin Oncol. 2001 Aug;28(4 Suppl 15):3-7. doi: 10.1016/s0093-7754(01)90148-4. PMID 11685722
- [Background] Picus J, Schultz M. Docetaxel (Taxotere) as monotherapy in the treatment of hormone-refractory prostate cancer: preliminary results. Semin Oncol. 1999 Oct;26(5 Suppl 17):14-8. PMID 10604263
- [Background] Hussain M, Smith DC, El-Rayes BF, Du W, Vaishampayan U, Fontana J, Sakr W, Wood D. Neoadjuvant docetaxel and estramustine chemotherapy in high-risk/locallyadvanced prostate cancer. Urology. 2003 Apr;61(4):774-80. doi: 10.1016/s0090-4295(02)02519-0. PMID 12670564
- [Background] Barton J, Blackledge G, Wakeling A. Growth factors and their receptors: new targets for prostate cancer therapy. Urology. 2001 Aug;58(2 Suppl 1):114-22. doi: 10.1016/s0090-4295(01)01253-5. PMID 11502465
- [Background] Sirotnak FM, Zakowski MF, Miller VA, Scher HI, Kris MG. Efficacy of cytotoxic agents against human tumor xenografts is markedly enhanced by coadministration of ZD1839 (Iressa), an inhibitor of EGFR tyrosine kinase. Clin Cancer Res. 2000 Dec;6(12):4885-92. PMID 11156248
- [Background] Oh WK, Kantoff PW. Treatment of locally advanced prostate cancer: is chemotherapy the next step? J Clin Oncol. 1999 Nov;17(11):3664-75. doi: 10.1200/JCO.1999.17.11.3664. PMID 10550165
- [Background] Simon R. Clinical trial designs for therapeutic cancer vaccines. Cancer Treat Res. 2005;123:339-50. doi: 10.1007/0-387-27545-2_14. PMID 16211877
- See also: Benaroya Research Institute at Virginia Mason is dedicated to discovering the causes of and cures for autoimmune and genetic diseases, to benefit patients with conditions such as diabetes, arthritis, and cancer. — http://www.benaroyaresearch.org